CLINICAL TRIAL: NCT00796133
Title: A Phase 2, Dose-finding, Cross-over Study to Evaluate the Effect of a NES/E2 Transdermal Gel Delivery on Ovulation Suppression in Normal Ovulating Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Population Council #427
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Ovulation
Keywords: NES/E2; transdermal gel delivery; contraception; ovulation; bleeding patterns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 0.5 ml of NES/E2 equaling 0.45 g and contains 1.5 mg NES/0.5 mg E2
  Interventions: Drug: NES/E2 gel
- 2 (Active Comparator): 1.0 ml of NES/E2 gel equaling 0.9 g and contains 3.0 mg NES/1.0 mg E2
  Interventions: Drug: NES/E2 gel
- 3 (Active Comparator): 1.5 ml of NES/E2 gel equaling 4.5 mg NES/1.5 mg E2
  Interventions: Drug: NES/E2 gel

INTERVENTIONS:
Drug: NES/E2 gel — Lowest effective dose of 3 formulations of the NES/E2 gel to ensure ovulation suppression (P<10nmol/L) in 90-95% of the cycles. The high dose will deliver 4.5mg of NES; the medium dose will deliver 3mg of NES, and a low dose of 1.5mg of NES. Based on a 10% absorption rate, 450 µg/d, 300 µg/d and 150 µg/d will be absorbed respectively. The doses of Estradiol will also be tailored to the 3 formulations.

SUMMARY:
This is a Phase 2, dose-finding, cross-over study for the purposes of evaluating the effect of a NES/E2 transdermal gel delivery on ovulation suppression in normal ovulating women.

ELIGIBILITY:
Inclusion Criteria:

* Woman is between 18 and 40 years of age
* Has intact uterus and ovaries
* Has regular menstrual cycles of 25-35 days duration
* Able to comply with the protocol, including frequent blood sampling, and lives within the catchment area of the clinic
* Understands the study procedures and agrees to participate in the study by giving written informed consent
* Able to use non-hormonal, double-barrier contraceptives (e.g. condoms and diaphragm) with every act of intercourse, or has been sterilized with tubal ligation, or only male partner has been sterilized with vasectomy
* Progesterone >10 nmol/L in at least one sample in the lead-in cycle

Exclusion Criteria:

* All contraindications to OC use including
* Thrombophlebitis or thromboembolic disorders
* Past history of deep vein thrombophlebitis or thromboembolic disorders
* Past or current cerebrovascular or coronary artery disease
* Known or suspected carcinoma of the breast
* Carcinoma of the endometrium or other known or suspected estrogen-dependent neoplasia
* Undiagnosed abnormal genital bleeding
* Cholestatic jaundice of pregnancy or jaundice with prior pill use
* Hepatic adenomas or carcinomas
* Woman has a history of headaches with focal neurological symptoms
* Known or suspected pregnancy
* Aged >35 and smoker
* BMI >29
* Positive urine pregnancy test at the screening or baseline visit
* Desired pregnancy within the duration of the study
* Known hypersensitivity to progestins
* Known hypersensitivity to estrogen
* Undiagnosed vaginal discharge or vaginal lesions or abnormalities
* In accordance with the Bethesda system of classification Women with a current abnormal Pap smear suggestive of high-grade pre cancerous lesion(s), including HGSIL, are excluded
* Women with LGSIL or ASCUS/high-risk HPV positive may participate if further evaluated with colposcopy and biopsy and no evidence of a lesion with a severity >CIN I is present and/or endocervical curettage is negative
* Women with a biopsy finding of CIN I should have follow up for this finding per standard of care; women are excluded if treatment is indicated In accordance with other Pap class systems
* Women with high grade dysplasia are excluded
* Women with low grade dysplasia or CIN I interpretation on Pap smear may participate based on investigator discretion in accordance with local standard of care
* Breastfeeding
* Cancer (past history of any carcinoma or sarcoma)
* History of a significant psychiatric disorder, including severe depression.
* Chronic or acute liver or renal disease
* Hypertension-- controlled by medication or defined by diastolic BP 85 mm Hg or systolic BP 135mm Hg after 15 minutes rest
* Dermatitis, psoriasis or other severe skin disorder
* Known or suspected alcoholism or drug abuse
* Clinically significant abnormalities of laboratory safety tests
* Chronic disease or history of illness that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject
* Woman is participating or has participated in another clinical study (involving an investigational drug) within one month prior to enrollment.
* Use of injectable contraceptives during the previous 3 months (e.g. cyclofem) or 9 months (e.g. DMPA)
* Use of oral contraceptives within the past 1 month
* Use of concomitant drugs that may interact with the study drugs

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Determine with ultrasound scan (USS) measures and serum progesterone (P) assessment the lowest effective dose of 3 formulations of the NES/E2 gel to ensure ovulation suppression (P<10nmol/L) in 90-95% of the cycles | Subjects will remain in the study for approximately 8 months

SECONDARY OUTCOMES:
Determine with USS and E2 serum levels the dose that can suppress follicle growth and replace estradiol at the physiological early follicular phase level | Subjects will remain in the study for approximately 8 months
Evaluate the correlation of NES and E2 serum levels with the percentage of ovulation suppression | Subjects will remain in the study for approximately 8 months
Evaluate the safety and tolerability of the formulations | Subjects will remain in the study for approximately 8 months

CONTACTS AND LOCATIONS:
Locations (3):
- Women's and Children's Hospital; LA County/USC Medical Center, Los Angeles, California, United States
- Instituto Chileno de Medicina Reproductiva, Santiago, Chile
- Profamilia, Santo Domingo, Dominican Republic

REFERENCES:
- [Derived] Brache V, Merkatz R, Kumar N, Jesam C, Sussman H, Hoskin E, Roberts K, Alami M, Taylor D, Jorge A, Croxatto H, Lorange E, Mishell DR, Sitruk-Ware R. A dose-finding, cross-over study to evaluate the effect of a Nestorone(R)/Estradiol transdermal gel delivery on ovulation suppression in normal ovulating women. Contraception. 2015 Oct;92(4):289-97. doi: 10.1016/j.contraception.2015.05.011. Epub 2015 May 29. PMID 26032952